CLINICAL TRIAL: NCT03850548
Title: Chronic Infections on Articular Prostheses With C. Acnes Diagnosed by Specific PCR : Descriptive Study of 6 Patients
Brief Title: Chronic Infections on Articular Prostheses With C. Acnes Diagnosed by Specific PCR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research assistant, Hospices Civils de Lyon
Other Study IDs: 18-031
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Bone and Joint Infection
Keywords: bone and joint infection; Propionibacterium acnes; Cutibacterium acnes
MeSH Terms: interventions — chloropentaamminerhodium(III)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prosthetic joint infection with Cutibacterium acnes: Chronic infections on articular prostheses with Cutibacterium acnes diagnosed by specific PCR
  Interventions: Other: Prosthetic joint infection with Cutibacterium acnes

INTERVENTIONS:
Other: Prosthetic joint infection with Cutibacterium acnes — patients having a prosthesis infection with C.acnes identified by specific PCR

SUMMARY:
Osteaoarticular infection due to C. acnes are known to be of late onset, causing chronic infection possibly pauci-symptomatic. Osteaoarticular infection due to C. acnes represents a diagnostic challenge, since C. acnes is slow and difficult to grow, and can also be considered a contaminant.A 16S universal PCR bacteriological diagnosis has been proposed but is lacking of sensitivity. A specific C. acnes PCR was developed in 2010, but is not used routinely.

ELIGIBILITY:
Inclusion Criteria:

* patients having had infection prothesis vith C. acnes identified by PCR

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had infection prothesis vith C. acnes identified by PCR and managed at the croix rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of diagnostic delay | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  time between surgery and detection of C. acnes by PCR

SECONDARY OUTCOMES:
rate of radiologic signs | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  prosthesis loosening or not
rate of duration of antibiotherapy | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  measures of duration of the antibiotherapy
rate of use of this diagnostic | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  descriptions of patients managed with this diagnostic

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Study Director — HCL
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided